CLINICAL TRIAL: NCT04210739
Title: Managment of Refractory Cases of Chronic Non Bacterial Prostatitis by TRUS Guided Injection of Betamethason
Brief Title: Chronic Non Bacterial Prostatitis: a Trial of TRUS Guided Injection of Betamethason
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abozamel, Doctor Lecturer in Urology department, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: chronic prostatitis
Record Dates: First submitted 2019-12-18; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Chronic Non Bacterial Prostatitis
MeSH Terms: interventions — betamethasone sodium phosphate

STUDY DESIGN:
Intervention Model Description: chronic non bacterial prostatitis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- trus guided betamethason injection arm (Experimental)
  Interventions: Drug: Betamethason Sodium Phosphate

INTERVENTIONS:
Drug: Betamethason Sodium Phosphate — Injection of betamethasone in chronic non bacterial prostatitis patients using Trans rectal Ultrasound

SUMMARY:
TRUS guided injection of long acting corticosteroids in chronic non bacterial prostatitis patients who failed to response to medical treamtment

DETAILED DESCRIPTION:
chronic non bacterial prostatitis is usually due to congestion combined with severe inflammatory process of the prostate, it is usually a recurrent bothersome problem, so patients who fail to response to classic medical treatment are expected to benefit from a strong anti inflammatory injection like betamethasone, which has strong anti inflammatory plus anti oedematous properties so limitation of this inflammatory process across the prostate is expected to relieve the patients symptoms

ELIGIBILITY:
Inclusion Criteria:

* chronic non bacterial prostatitis who failed medical treatment

Exclusion Criteria:

* chronic bacterial prostatitis patients

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Comparing IPSS before and after injection. | evaluation over 3 months after injection
  Questionnaire comparing IPSS (international prostatic symptom score) before and after injection